

## NFORMED CONSENT

Study title:

## Evaluation of the Efficacy of Chlorhexidine Use During the First Trimester as a Regulator of Vaginal Microbiota in Reducing Preterm Birth

- I, (name and surname).
- -I have read the information sheet given to me.
- -I have been able to ask questions about the study.
- -I have received sufficient information about the study.
- -I have spoken to: (Dr. Morales Roselló, Dr. Loscalzo).
- -I understand that my participation is voluntary.
- -I will receive a signed and dated copy of this informed consent document.

I understand that I can withdraw from the study:

- -1° Whenever I want
- -2° Without having to give explanations.
- -3° Without any repercussions on my medical care.

| I freely give my agreement to participate in | n the study. |
|---|---|
| | José Morsles Rosello |
| Participant's Signature Name: Date:// | Researcher's signature<br>Name: Dr.José Morales Roselló<br>Date:// |
| I wish to be informed of information derive ☐ YES ☐ NO | ed from the research that may be relevant to my health: |